CLINICAL TRIAL: NCT02654249
Title: Prospective Multicenter Randomized Trial About Transanal Hemorrhoidal Dearterialization With Mucopexy (THD) Versus Ligasure Hemorrhoidectomy for Grade III and IV Hemorrhoids
Brief Title: Prospective Randomized Trial About THD Versus Ligasure Hemorrhoidectomy for Grade III and IV Hemorrhoids
Acronym: THD-LIGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Sebastiano Biondo, MD, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THD_LIGA_RCT
Record Dates: First submitted 2015-12-13; First posted 2016-01-13 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids grade III and IV; transanal hemorrhoidal dearterialization; hemorroidectomy; THD; LigaSure
MeSH Terms: conditions — Hemorrhoids | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- THD and mucopexy (Other): Patients will undergo to transanal hemorrhoidal dearterialization with mucopexy (THD)‪ under generla anesthesia.
  Interventions: Device: Transanal hemorrhoidal dearterialization + mucopexy (THD).; Device: THD anoscope and doppler
- Ligasure hemorroidectomy (Active Comparator): Patients will undergo to Ligasure™ hemorroidectomy under generla anesthesia.
  Interventions: Procedure: Ligasure™ hemorrhoidectomy; Device: Ligasure Vessel Sealing

INTERVENTIONS:
Device: Transanal hemorrhoidal dearterialization + mucopexy (THD). — Using an anoscope combined with a Doppler transducer the hemorrhoidal arteries are identified and ligated to decrease the blood flow to the hemorrhoidal plexus. In order to reduce hemorroidal prolapse a mucopexy is performed.
  Arms: THD and mucopexy
Procedure: Ligasure™ hemorrhoidectomy — Excisional hemorroidectomy performed with Ligasure™
  Arms: Ligasure hemorroidectomy
Device: THD anoscope and doppler — An dedicated anoscope with an incorporated doppler probe sold by THD Lab S.p.A will be used for the THD procedure
  Arms: THD and mucopexy
Device: Ligasure Vessel Sealing — A curved, small jaw, open sealer/divider sold by Covidien/medtronic will be used for the Ligasure™ hemorrhoidectomy
  Arms: Ligasure hemorroidectomy

SUMMARY:
The study evaluates postoperative pain, morbidity, recurrence and quality of life, comparing two different strategies in the treatment of grade III and IV hemorrhoids: transanal hemorrhoidal dearterialization with mucopexy (THD) versus hemorrhoidectomy by Ligasure™.

DETAILED DESCRIPTION:
Transanal hemorrhoidal dearterialization (THD)‪ uses a specially developed anoscope combined with a Doppler transducer to identify the hemorrhoidal arteries. A suture ligation is performed to effectively decrease the blood flow to the hemorrhoidal plexus. In case of redundant prolapse, the prolapsed mucosa is lifted (mucopexy). THD procedure is performed without any incisions or removal of the hemorrhoidal tissue and moreover the suture line is above the dentate line, so post-operative pain and morbidities seem to be minimized in these patients. This technique differs from Ligasure hemorrhoidectomy, which focuses on excising the hemorrhoidal tissue.

This prospective, randomized, multicenter and controlled trial compares post-operative pain, morbidities, quality of life, fecal incontinence and recurrence rate in patients treated for grade III and IV hemorrhoids with THD with mucopexy versus Ligasure hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade III and IV hemorrhoids according to Goligher classification
* Patients ASA I, II or III and adequate hematological, renal and hepatic function
* Patients who signed informed consent

Exclusion Criteria:

* Altered cognitive state that prevents collaboration in the study or patients who can neither read nor write
* Fecal incontinence
* Anal sphincter lesions
* Recurrent hemorrhoids after previous surgical tratment
* Previous anorectal surgery except banding, botulinum toxin injection and thrombectomy for hemorrhoid thrombosis
* Injection sclerotherapy during the last five years
* Concomitant anorectal disease (anal fistula, anal fissure, anal stenosis, rectocele, enterocele, anal condilomatosis).
* Concomitant diagnosis of functional pelvic floor disease, inflammatory bowel disease and previous pelvic radiotherapy
* Concomitant diagnosis of colorectal neoplasia or other neoplasia
* Patients ASA IV, V
* NSAIDs, Paracetamol, Tramadol, Metamizol and Petidine allergy
* Coagulation disorders
* Pregnancy and lactation
* Rejection of the patient to sign the consent form.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | within the first 30 days after surgery
  Post-operative pain by simple verbal numerical scale (0-10), the Andersen scale (0-5) and the taken pain medicacions will be recorded by the patients on a specific book during the first thirty days after surgery.

SECONDARY OUTCOMES:
Quality of life | At 1 month and at 1 and 2 years after surgery
  Quality of life by Short Form 12 (SF-12) Questionnaire
Specific disabilities (fecal incontinence and costipation) | At the day 15, 30 and at 1 and 2 years after surgery
  Fecal incontinence by Vaizey Score and need of laxatives. Anorecatal manometry and endoanal ultrasonography will be performed two month after surgery.
Post-operative morbidity | within the first 30 days after surgery
  Dindo classification of complicacions will be used
Hemorrhoid recurrence | At 1 and 2 years after surgery
  rectal bleeding, anal pain, mucosal prolaps will be invastigated one year after hemorroidectomy. Needing of further surgery for hemorrhoids recurrence will be recorded
Satisfaction after surgery | At the day 15, 30 and at 1 and 2 years after surgery
  A scale of 0-3 (0, not satisfied; 1 few satisfied, 2 satisfied, 3, very satisfied) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, MD, PhD, Principal Investigator — Bellvitge University Hospital
Locations (10):
- Spain (10):
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona
  - Galdakano Usansolo Hospital, Bizkaia, Basque Country
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Comarcal de Valdeorras, O Barco de Valdeorras, Ourense
  - Hospital Universitario de la Ribera, Alzira, Valencia
  - Valle d'Hebron University Hospital, Barcelona
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario de La Princesa, Madrid
  - Fundación Jimenez Diaz, Madrid
  - Hospital La Paz, Madrid

REFERENCES:
- [Derived] Trenti L, Biondo S, Espin-Basany E, Barrios O, Sanchez-Garcia JL, Landaluce-Olavarria A, Bermejo-Marcos E, Garcia-Martinez MT, Alias Jimenez D, Jimenez F, Alonso A, Manso MB, Kreisler E; THDLIGA-RCT Study Group. Transanal Hemorrhoidal Dearterialization With Mucopexy Versus Vessel-Sealing Device Hemorrhoidectomy for Grade III to IV Hemorrhoids: Long-term Outcomes From the THDLIGA Randomized Controlled Trial. Dis Colon Rectum. 2023 Aug 1;66(8):e818-e825. doi: 10.1097/DCR.0000000000002272. Epub 2022 Mar 1. PMID 35239526
- [Derived] Trenti L, Biondo S, Kreisler Moreno E, Sanchez-Garcia JL, Espin-Basany E, Landaluce-Olavarria A, Bermejo-Marcos E, Garcia-Martinez MT, Alias Jimenez D, Jimenez F, Alonso A, Manso MB; THDLIGA-RCT Study Group. Short-term Outcomes of Transanal Hemorrhoidal Dearterialization With Mucopexy Versus Vessel-Sealing Device Hemorrhoidectomy for Grade III to IV Hemorrhoids: A Prospective Randomized Multicenter Trial. Dis Colon Rectum. 2019 Aug;62(8):988-996. doi: 10.1097/DCR.0000000000001362. PMID 30807456